CLINICAL TRIAL: NCT00385385
Title: Randomized Evaluation of Short-Term Rifalazil Treatment on Carotid Atherosclerosis and Intima Media Thickness
Brief Title: RESTORE-IT-Study of Rifalazil in Chlamydia Pneumoniae Seropositive Patients With a History of Atherosclerotic Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ActivBiotics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ABI-1648-026
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Coronary Artery Disease; Cerebrovascular Disease; Peripheral Vascular Disease
MeSH Terms: conditions — Coronary Artery Disease; Cerebrovascular Disorders; Peripheral Vascular Diseases | interventions — KRM 1648

INTERVENTIONS:
Drug: Rifalazil

SUMMARY:
The objective of this study is to evaluate an antibiotic therapy called Rifalazil to determine its effect on hardening of the carotid arteries.

DETAILED DESCRIPTION:
To evaluate the effect of treatment with rifalazil versus placebo taken once weekly for 12 weeks on carotid atherosclerotic disease progression in patients who test positive for Chlamydia pneumoniae. Measurements of the carotid artery wall (intima-media thickness) and plaque characteristics will be evaluated with high-resolution magnetic resonance imaging (MRI) and carotid ultrasound. at Baseline and at 6,12 and 18 months following initiation of drug treatment in Chlamydia pneumoniae seropositive patients with a history of atherosclerotic disease. Biomarkers will be collected throughout the study. Safety will be evaluated by the collection and analysis of laboratory parameters, vital signs, electrocardiograms, physical examination and adverse events. Seventy two patients will be enrolled in this study. There will be a total of approximately 7-9 visits which will occur over an 18 month period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 50 and 85 years of age.
* Patient has seropositive evidence of C. pneumoniae defined by IgG antibody titers ≥ 1:128 on microimmunofluorescence assay.
* The patient meets at least one of the following criteria:

  1. Diagnosis of PAD: i. Ankle-brachial index (ABI) of <0.90 at rest in either leg, or toe brachial index of < 0.7 if ankle pressure is calcified. ii. Known PAD on the basis of history or symptoms of intermittent claudication, prior endovascular or surgical revascularization.
  2. Known large vessel (non-cardioembolic) cerebrovascular event (stroke or TIA) within the last three years or carotid stenosis of >40% and ≤ 80% by Doppler ultrasound or asymptomatic carotid artery disease defined by a total plaque area >100 mm2and carotid stenosis of ≤ 80%by Doppler ultrasound.
  3. Known coronary artery disease on the basis of an exercise tolerance test positive for myocardial ischemia, or history of a prior myocardial infarction (greater than 6 months), or prior percutaneous coronary intervention and/or surgical revascularization (greater that 6 months).
* Patient has a maximal IMT measurement by ultrasound in either the left or right common carotid artery of ≥ 0.70 mm and at least one or more echogenic carotid plaques detectable in either the right or left side of the carotid artery.
* Patient is able to undergo magnetic resonance (MR) examination and MR baseline images obtained are of suitable image quality for analysis.
* If patient is taking cilostazol, pentoxifylline, or other approved drugs for the treatment of PAD and/or intermittent claudication or taking a statin, patient has to be on the medication for at least 6 months prior to Screening.
* Patients who have recently discontinued medications for PAD and/or intermittent claudication or statin must "wash-out" for at least one month prior to screening.
* Male and female patients must agree to use an effective form of birth control throughout the study period.

Exclusion Criteria:

* The patient lacks evidence of intermediate or advanced carotid atherosclerotic lesions or has heavily calcified plaque or poor image quality of their carotid arteries as determined by the MRI lab.
* Patient has critical limb ischemia as evidenced by ischemic rest pain, ulceration, or gangrene.
* Patient has new, previously unrecognized clinically significant electrocardiogram (ECG) abnormalities.
* Patient has liver function tests > 3.0 times the upper limit of normal, serum creatinine > 1.8 mg/dL for females and >2.0 mg/dL for males and a eGFR value <30 mL/min/1.73 m2. Enrollment of patients with eGFR values of between 30 and 59 mL/min/1.73 m2 will be left to the discretion of the investigator. Patients with abnormal laboratory values which are deemed clinically significant by the investigator will not be enrolled.
* Patient has had a recent (< 6 months) coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), carotid endarterectomy (CEA), carotid artery stent, or lower extremity revascularization/amputation.
* Patient plans for surgical/endovascular intervention for carotid and/or coronary during the course of the study.
* Patient has or being evaluated or treated for tuberculosis. Patients who were treated previously for tuberculosis but presently have inactive disease may be included.
* Patient has a chest x-ray obtained within the last month that is consistent with possible tuberculosis.
* Patient has a history of malignant neoplasm within the previous 5 years (except curable non-melanoma skin malignancies).
* Patient has a known immunodeficient state or is being treated with immunosuppressive drugs including high-dose steroids or cyclosporine.
* Patient has an active infection requiring systemic or oral antibiotics. Patients with prior infection must have discontinued such treatments at least 14 days prior to administration of investigational agent.
* Patient has an uncontrolled, unstable or recently diagnosed autoimmune disease, including but not limited to systemic lupus, inflammatory bowel disease, sarcoidosis, rheumatoid arthritis, or psoriasis.
* Patient has a recent history of alcohol abuse, illicit drug use or drug abuse or significant mental illness.
* Patient has a known or suspected allergy to the study medication(s) or class of study medication (rifamycins).
* Patient chronically uses antibacterials or has previously received rifalazil.
* Patient has a known or suspected allergy to MRI contrast agents (e.g., gadolinium) and/or has any medical or physical condition that would prevent them from receiving a gadolinium-based contrast agent or an MRI examination.
* Patient has participated in any clinical trial of an investigational drug, device, or medical procedure within 30 days prior to Baseline of the study.
* Patient is enrolled or plans to enroll in another clinical drug or device/interventional trial during this study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-10; Study Completion 2008-09

PRIMARY OUTCOMES:
To evaluate the treatment with Rifalazil versus placebo on high-resolution magnetic resonance imaging (MRI) determined by the normalized wall index (NWI) over a segment of the carotid artery at Day 180.
NWI is defined as the wall area (WA) over the length of the arterial segment studied divided by the sum of the wall area plus the lumen area (LA) over the length of the arterial segment studied [NWI = WA / (WA + LA)].

SECONDARY OUTCOMES:
To evaluate the effect of rifalazil versus placebo on carotid intima media thickness (IMT), and carotid plaque composition by ultrasound and MRI and to determine the overall safety of a 12 week regimen of rifalazil administered once weekly.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Thoracic & Cardiovascular Healthcare Foundation, Lansing, Michigan
  - St. Francis Hospital, Roslyn, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Baylor College of Medicine, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
- Robarts Research Institute, London, Ontario, Canada